CLINICAL TRIAL: NCT04243824
Title: The Evaluation of Ga-68 MAA Distribution in Prostatic Artery Embolization Patients
Brief Title: Ga-68 MAA Distribution in PAE Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: BTG International Inc. (Other); Embolx, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-2669
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All enrolled study participants will receive Ga-68MAA and PET/MRI scan.
  Interventions: Drug: Gallium 68 Macro-aggregated albumin

INTERVENTIONS:
Drug: Gallium 68 Macro-aggregated albumin — The radiotracer, Ga-68 MAA, will be administered prior to PET/MRI scan.
  Other Names: radiotracer

SUMMARY:
Purpose: The purpose of this study is to evaluate Ga-68 MAA distribution on PET/MRI after injection into the prostatic arteries in patients without prostate cancer who are being treated with prostate artery embolization for benign prostatic hyperplasia.

Participants: Study subjects will be 5 men scheduled to undergo the PAE procedure at UNC Hospital for benign prostatic hyperplasia.

Procedures (methods): Study subjects will undergo PAE using the standard technique. Prior to embolization of the prostatic artery with the bland embolic agent, Ga-68 MAA will be injected. Standard departmental radiation protection procedures will be followed. After the PAE procedure is complete, the patient will be transported to the UNC Biomedical Research Imaging Center to undergo PET/MRI.

DETAILED DESCRIPTION:
This study is an initial proof of concept evaluation to determine the feasibility of using Y-90 radioembolization performed using the Sniper balloon occlusion microcatheter to treat localized prostate cancer. This will be performed by evaluating Ga-68 MAA distribution on PET/MRI after injection into the prostatic arteries in patients without prostate cancer who are being treated with prostate artery embolization for benign prostatic hyperplasia. The distribution of the radiotracer activity within the prostate and any activity in adjacent organs will be determined for when the tracer is injected into the central prostatic arteries.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age > 40
* Prostate gland >50 grams as measured by pre-procedural CTA
* Have previously taken BPH medication for 6 months without desired improvement of LUTS or has started medication and stopped due to unwanted side effects
* Moderate to severe LUTS as defined by IPSS score >18
* Peak urine flow rate (Qmax) <12 mL/sec
* Capable of giving informed consent
* Life expectancy greater than 1 year

Exclusion Criteria:

* Severe vascular disease
* Uncontrolled diabetes mellitus
* Immunosuppression
* Unable to lie flat, still or tolerate a PET/MRI scan.
* Neurogenic bladder and/or sphincter abnormalities secondary to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes, etc.
* Complete urinary retention
* Impaired kidney function (serum creatinine level > 1.8 mg/dl or a glomerular filtration rate < 60 as approximated using serum creatinine levels) unless anuric and on dialysis.
* Confirmed or suspected bladder cancer
* Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology
* Ongoing urogenital infection
* Previous pelvic radiation or radical pelvic surgery
* Confirmed or suspected malignancy of the prostate based on DRE, TRUS or PSA (> 10 ng/mL or > 4.0 ng/mL and < 10 ng/mL with free PSA < 25% of total PSA without a negative biopsy).
* Uncorrectable coagulopathy including INR > 1.5 or platelets < 50,000
* Contrast hypersensitivity refractory to standard medications (antihistamines, steroids)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender is based on the anatomical gender assigned at birth. Patients must have a prostate in order to enroll in this study.
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Ga-68 MAA radiotracer activity within adjacent organs | Upon completion of all study image data collection for all participants [approximately 1 year]
  The mean radiotracer levels within adjacent organs in the target population of patients will be estimated in the sample of N=5 patients, along with standard errors, and 95% confidence intervals.

SECONDARY OUTCOMES:
Ga-68 MAA radiotracer activity within the prostate gland | Upon completion of all study image data collection for all participants [approximately 1 year after study start]
  The mean radiotracer amounts within the central and peripheral prostate gland in the target population of patients will be estimated in the sample of N=5 patients, along with standard errors, and 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Stewart, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.